CLINICAL TRIAL: NCT04984057
Title: Optimal Dose of Surfactant for Preterm Infants With Respiratory Distress Syndrome(RDS)
Brief Title: Optimal Dose of Surfactant for Preterm Infants With Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Director, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Surfactant dose
Record Dates: First submitted 2021-07-24; First posted 2021-07-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Distress Syndrome, Newborn; Patent Ductus Arteriosus; Bronchopulmonary Dysplasia; Preterm
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Ductus Arteriosus, Patent; Bronchopulmonary Dysplasia; Premature Birth | interventions — acetylamino propylidene diphosphonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS is stopped when the pressure is equal between bPDA and aPDA (Experimental): PS is given and stopped when the pressure is equal between bPDA and aPDA. the pressure is measured using ultrasound
  Interventions: Drug: PS is stopped when the pressure is equal between bPDA and aPDA.
- PS is given according to the 2019 European RDS management guideline (Active Comparator): PS is given according to the 2019 European RDS management guideline
  Interventions: Drug: PS is given according to the 2019 European RDS management guideline

INTERVENTIONS:
Drug: PS is stopped when the pressure is equal between bPDA and aPDA. — PS is given and stopped when the pressure is equal between bPDA and aPDA. the pressure is measured using ultrasound
  Arms: PS is stopped when the pressure is equal between bPDA and aPDA
Drug: PS is given according to the 2019 European RDS management guideline — PS is given according to the 2019 European RDS management guideline
  Arms: PS is given according to the 2019 European RDS management guideline

SUMMARY:
In preterm infants with neonatal respiratory distress syndrome (RDS), exogenous pulmonary surfactant(PS) replacement therapy is one of the most important therapeutic breakthrough to reduce neonatal incidences of bronchopulmonary dysplasia(BPD) and/or death. But not all preterm infants with RDS can be beneficial. Otherwise, the international neonatal acute RDS (NARDS) collaborative group provides the first consensus definition for NARDS in 2017. And whether or not PS being beneficial in preterm infants with NARDS remains unknown.

DETAILED DESCRIPTION:
To date, the optimal dose of PS is inconsistent, although the recommended dose of PS is given in the 2019 update guideline. PS is not recommended to adult and pediatric ARDS. Systematic review indicates that PS does not reduce the incidences of BPD and death in infants with meconium aspiration syndrome(MAS, a subtype of NARDS). A reasonable speculation is that preterm infants with NARDS do not benefit from PS. And the speculation can explain why not all preterm infants with RDS can be beneficial from PS. In the era of pre-NARDS, the preterm infants fulfilling the definition of NARDS may have been considered as RDS in the first three days after birth.

Meantime, the dose of PS given to infants with NARDS remains unknown. the aim of the present study is to assess the optimal dose of PS. the control group: PS is given according to the European RDS management guideline in 2019 edition. The study group: PS is stopped when the pressure is equal between before patent ductus arteriosus(bPDA) and after PDA(aPDA). the primary outcomes are the closure rate of PDA within 7 days, the incidence of BPD and/or death.

ELIGIBILITY:
Inclusion Criteria:

* gestation age less than or equal to 32 weeks
* PS is needed

Exclusion Criteria:

* main congenital abnormalities
* parents' refusal or quit

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the size of PDA | within 7 days after birth
  the size of PDA is zero
BPD and/or death | at 36 week's gestational age
  the BPD and/or death is diagnosed when the included infants remain needing oxygen at 36 week's gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, China